CLINICAL TRIAL: NCT06486545
Title: Liposomal Irinotecan Combined With Albumin-bound Paclitaxel for Second-line Treatment of Advanced Gastric Cancer: a Single-arm, Single-center Clinical Study
Brief Title: Liposomal Irinotecan Combination Regimen for Second-line Treatment of Advanced Gastric Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hunan Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: nal-IRI-GC-01
Record Dates: First submitted 2024-06-21; First posted 2024-07-03 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-06

CONDITIONS: Advanced Gastric Cancer
Keywords: Gastric cancer and gastroesophageal junction adenocarcinoma; Liposomal irinotecan; Albumin-paclitaxel; Second-line treatment; Dose escalation
MeSH Terms: conditions — Stomach Neoplasms | interventions — Injections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Liposomal irinotecan + Albumin-paclitaxel (Experimental): Liposomal irinotecan, intravenous infusion 90min, d1:
  Grade 1:50mg/m2； Grade 2:60mg/m2； Grade 3:70mg/m2；
  Albumin-paclitaxel, 150mg/m2, intravenous infusion, d1
  Interventions: Drug: Irinotecan Hydrochloride Liposome Injection；Paclitaxel For Injection (Albumin Bound)

INTERVENTIONS:
Drug: Irinotecan Hydrochloride Liposome Injection；Paclitaxel For Injection (Albumin Bound) — Liposomal irinotecan, intravenous infusion 90min, d1:
  Grade 1:50mg/m2； Grade 2:60mg/m2； Grade 3:70mg/m2；
  Albumin-paclitaxel, 150mg/m2, intravenous infusion, d1
  DLT was observed for 2 weeks (the first cycle). The same subject received only one dose of liposomal irinotecan during the study. If the patient volunteers and the investigator determines that the benefits of continuing the original regimen outweigh the risks, the subject may continue to receive treatment for metastatic disease. The drug was repeated every 2 weeks for up to 6 cycles, and the albumin paclitaxel or liposomal irinotecan were withdrawn according to the patient's adverse reactions and physical status, and the remaining single-agent maintenance therapy was performed. Until there is a possibility of surgery, disease progression, intolerable toxicity or the patient withdraws informed consent (whichever comes first).

SUMMARY:
Liposomal irinotecan, intravenous infusion 90min, d1:

Grade 1:50mg/m2 Grade 2:60mg/m2 Grade 3:70mg/m2 Albumin-paclitaxel, 150mg/m2, intravenous infusion, d1 DLT was observed for 2 weeks (the first cycle). The same subject received only one dose of liposomal irinotecan during the study. All subjects underwent protocol-mandated examinations during treatment to observe safety and initial efficacy. If the patient volunteers and the investigator determines that the benefits of continuing the original regimen outweigh the risks, the subject may continue to receive treatment for metastatic disease. The drug was repeated every 2 weeks for up to 6 cycles, and the albumin paclitaxel or liposomal irinotecan were withdrawn according to the patient's adverse reactions and physical status, and the remaining single-agent maintenance therapy was performed. Until there is a possibility of surgery, disease progression, intolerable toxicity or the patient withdraws informed consent (whichever comes first).

DETAILED DESCRIPTION:
This is a single-arm, single-center clinical study to evaluate the efficacy and safety of liposomal irinotecan combined with albumin paclitaxel regimen for second-line treatment of advanced gastric cancer. Using a "3+3" study design, 9 to 18 eligible patients with unresectable or locally advanced gastric cancer and gastroesophageal junction adenocarcinoma will receive liposomal irinotecan + albumin paclitaxel combination therapy.

Three dose groups of liposomal irinotecan 50mg/m2, 60 mg/m2 and 70 mg/m2 were preset, and a fixed dose of albumin paclitaxel (150mg/m2, intravenous infusion, d1) was administered for one cycle. The dose of liposomal irinotecan was gradually increased from the low-dose group to the high-dose group, and DLT was observed for 2 weeks (the first cycle). The same subject received only one dose of liposomal irinotecan during the study. All subjects underwent protocol-mandated examinations during treatment to observe safety and initial efficacy. If the patient volunteers and the investigator determines that the benefits of continuing the original regimen outweigh the risks, the subject may continue to receive treatment for metastatic disease. The drug was repeated every 2 weeks for up to 6 cycles, and the albumin paclitaxel or liposomal irinotecan were withdrawn according to the patient's adverse reactions and physical status, and the remaining single-agent maintenance therapy was performed. Until there is a possibility of surgery, disease progression, intolerable toxicity or the patient withdraws informed consent (whichever comes first).

Main study indicators: Maximum tolerated dose (MTD) of liposomal irinotecan in the combination regimen; Secondary study measures: dose-limiting toxicity (DLT) of liposomal irinotecan, objective response rate (ORR), disease control rate (DCR), progression-free survival (PFS), and overall survival (OS) .

ELIGIBILITY:
Inclusion Criteria:

* Patients fully understand the study, voluntarily participate and sign an informed consent form (ICF)
* Age ≥18 years
* The expected survival time is ≥3 months
* Patients with histologically or pathologically confirmed unresectable or locally advanced gastric cancer and gastro-oesophageal junction adenocarcinoma
* Patients who have progressed after previous first-line treatment based on fluorouracil
* HER-2+ is known to have been previously trastuzumab or HER-2 negative
* According to RECIST1.1 criteria, the patient had at least one measurable target lesion
* Eastern Cooperative Oncology Group（ECOG）Physical status score: 0-2
* Absolute neutrophil count (ANC) ≥1.5×10^9/L, platelets ≥100×10^9/L, and hemoglobin ≥90 g/L
* Serum creatinine ≤1.5 times the upper limit of normal value; AST and ALT ≤2.5 times the upper limit of normal (≤5 times the upper limit of normal for patients with liver invasion); Total bilirubin ≤1.5 times the upper limit of normal (≤3 times the upper limit of normal for patients with liver invasion)
* There are no contraindications for the use of liposomal irinotecan and albumin paclitaxel
* Women of childbearing age must have had a pregnancy test (serological) negative within 7 days prior to enrollment and be willing to use an appropriate method of contraception during the trial
* Agree to provide histological samples

Exclusion Criteria:

* Allergic reaction to any investigational drug or its ingredients
* Patients with relapse within 6 months after previous first-line treatment with paclitaxel
* The investigational agent was a CYP3A4 strong inducer within 2 weeks prior to initial administration, or a CYP3A4 strong depressant or UGT1A1 strong depressant within 1 week
* Uncontrolled systemic diseases (e.g. advanced infections, uncontrolled hypertension, diabetes, etc.)
* Imaging confirmed intestinal obstruction
* It has uncontrollable ascites, abdominal infection and pyloric obstruction
* Hepatitis B, hepatitis C active infection (hepatitis B surface antigen positive and hepatitis B DNA more than 1x103 copies /mL; more than 1x103 copies /mL of HCV RNA)
* Human immunodeficiency virus (HIV) infection (HIV antibody positive)
* Previous or current co-occurrence of other malignancies (in addition to non-melanoma basal cell carcinoma of the skin that is effectively controlled, breast/cervical carcinoma in situ, and other malignancies that have been effectively controlled without treatment within the past five years)
* Pregnant and lactating women and patients of childbearing age who do not want to use contraception
* The investigators determined that patients were not suitable to participate in this study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2024-08-25 (Estimated); Primary Completion 2025-07-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose | From the recorded first dose of Liposomal irinotecan to 4 weeks after the recorded last dose of Liposomal irinotecan.
  To estimate the maximum tolerated dose of liposomal irinotecan in the combination regimen based on dose-limiting toxicity

SECONDARY OUTCOMES:
Dose-limiting Toxicity (DLT) of liposomal irinotecan | From the recorded first dose of Liposomal irinotecan to 4 weeks after the recorded last dose of Liposomal irinotecan.
  One or more adverse events that occurred during the DLT observation period related to the investigational drug (including definitely related, likely related, possibly related) (meeting the DLT criteria)
Objective response rate | Data obtained up until progression, or the last evaluable assessment in the absence of progression, will be assessed up to 2 years.
  Per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) using lnvestigator assessments, is defined as the number (%) of paients of Complete Response or Partial Response, will be assessed up to 2 years.
Disease control rate | Data obtained up until progression, or the last evaluable assessment in the absence of progression, will be assessed up to 2 years.
  The percentage of subiects of Complete Response (CR) or Parial Response (PR) or Stable Disease (SD) by Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) as assessed by the investigator, will be assessed up to 2 years.
Progression-free survival | Progression-free survival (PFS) analysis based on investigator assessment per RECIST 1.1, and will be assessed up to 2 years.
  Progression-free survival (PFS) is defined as the time from first dose of Liposomal irinotecan recorded until the date of disease progression based on investigator assessment.
Overall survival | The time from beginning of Liposomal irinotecan treatment until death due to any cause and will be assessed up to 3 years.
  Overall survival is defined as the time from begining of Liposomal irinotecan treatment until death due to any cause and wil be assessed up to 3 years.

CONTACTS AND LOCATIONS:
Overall Officials: Liu zhenyang, Doctor, Principal Investigator — Hunan Cancer Hospital

IPD SHARING:
Plan to Share IPD: Yes
Information about this clinical study will be posted on the Chinese Clinical Trials Registry or clinicaltrials.gov website
Supporting Information: Study Protocol, ICF